CLINICAL TRIAL: NCT04419467
Title: A Phase 2a, Double-blind, Randomized, Placebo-controlled, Proof of Concept Study of Vascular Endothelial Growth Factor (VEGF)-B Blockade With the Monoclonal Antibody CSL346 in Subjects With Diabetic Kidney Disease
Brief Title: Vascular Endothelial Growth Factor-B (VEGF-B) Blockade With the Monoclonal Antibody CSL346 in Subjects With Diabetic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL346_2001
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Kidney Disease (DKD)
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CSL346 (low dose) (Experimental): Administered as a single intravenous (IV) loading dose followed by subcutaneous (SC) infusions
  Interventions: Biological: CSL346
- CSL346 (high dose) (Experimental): Administered as a single intravenous (IV) loading dose followed by subcutaneous (SC) infusions
  Interventions: Biological: CSL346
- Placebo (Placebo Comparator): Administered as a single IV loading dose followed by SC infusions
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CSL346 — VEGF-B antagonist monoclonal antibody
  Arms: CSL346 (high dose); CSL346 (low dose)
Drug: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
This phase 2a, double-blind, randomized, placebo-controlled study will assess the efficacy, safety, tolerability, and pharmacokinetics (PK), of repeat doses of CSL346 in subjects with diabetic kidney disease (DKD) and albuminuria receiving standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 25 years of age with a diagnosis of type 2 diabetes mellitus (T2DM)
* Urinary ACR ≥ 150 mg/g
* eGFR > 20 mL/min/1.73m2
* Glycosylated HbA1c < 12%

Exclusion Criteria:

* Current diagnosis of type 1 diabetes mellitus
* History of acute kidney injury or chronic dialysis/renal transplant
* Uncontrolled hypertension or class III / IV heart failure
* Left ventricular ejection fraction < 50% by echocardiogram
* Troponin-I > the upper reference limit
* b-type natriuretic peptide > 200 pg/mL
* ALT > 2x the upper limit of normal

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (37):
- United States (22):
  - California Kidney Specialists (CKS) - Citrus Office, Covina, California
  - Valley Research - Fresno, Fresno, California
  - Torrance Clinical Research (TCR) - Lomita, Lomita, California
  - Renal Medical Associate/NARI, Lynwood, California
  - Amicis Research Center, Northridge, California
  - California Medical Research Associates, Inc, Northridge, California
  - Riverside Nephrology Group, Riverside, California
  - West Orange Endocrinology, Ocoee, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Omega Clinical Research, Metairie, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Renal and Transplant Associates, Springfield, Massachusetts
  - University of Missouri Health System, Columbia, Missouri
  - Palm Medical Group, LLC - Las Vegas, Las Vegas, Nevada
  - Center for Thyroid & Parathyroid Disorders, Staten Island, New York
  - Physicians East, P.A. - Endocrinology, Greenville, North Carolina
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - Juno Research, L.L.C., Houston, Texas
  - The Endocrine Center, Houston, Texas
  - Renal Associates, P.A. - San Antonio, San Antonio, Texas
  - Primary Care Providers of Texas, San Antonio, Texas
  - Diabetes and Metabolism Specialists (DMS) - San Antonio, San Antonio, Texas
- Australia (6):
  - Hunter Diabetes Centre - The AIM Centre, Merewether, New South Wales
  - St Vincent's Hospital, Fitzroy, Victoria
  - The Austin Hospital, Heidelberg, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Lyell McEwin Hospital, Elizabeth Vale
- 1240130 - University Health Network, Toronto, Ontario, Canada
- Israel (2):
  - 3760045 - Kaplan Medical Center, Rehovot
  - 3760044 - Tel Aviv Sourasky Medical Center, Tel Aviv
- New Zealand (4):
  - Middlemore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Lipid and Diabetes Research Group, Christchurch
  - Endocrine Associates - Wellington, Wellington
- Puerto Rico (2):
  - Fundación de Investigación, San Juan
  - University of Puerto Rico - Puerto Rico Clinical and TRC, San Juan

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.

REFERENCES:
- [Derived] Cooper M, Cherney DZI, Greene TH, Heerspink HJL, Jardine M, Lewis JB, Wong MG, Baquero E, Heise M, Jochems J, Lanchoney D, Liss C, Reiser D, Scotney P, Velkoska E, Dwyer JP. Vascular Endothelial Growth Factor-B Blockade with CSL346 in Diabetic Kidney Disease: A Phase 2A Randomized Controlled Trial. J Am Soc Nephrol. 2024 Nov 1;35(11):1546-1557. doi: 10.1681/ASN.0000000000000438. Epub 2024 Aug 16. PMID 39150859

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study centers in Australia, Canada, Israel, New Zealand, Puerto Rico and the United States.
Pre-assignment Details: A total of 327 participants were screened, of which 114 participants met the eligibility criteria, completed the Lead-in Period and were randomized to receive CSL346 (low dose), CSL346 (high dose), or Placebo.
Period: Overall Study
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose) | Placebo
Started | 29 | 29 | 56
Completed | 27 | 26 | 47
Not Completed | 2 | 3 | 9
Not completed — Not treated with IP | 0 | 0 | 2
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Pandemic related | 0 | 0 | 1
Not completed — Reason not known | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose) | Placebo | Total
Number analyzed (Participants) | 29 | 29 | 56 | 114
Age, Continuous [Median (Full Range); unit: Years] | 62.0 [37 to 78] | 61.0 [39 to 84] | 63.0 [32 to 85] | 62.0 [32 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 11 | 28
  Male | 19 | 22 | 45 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 19 | 36
  Not Hispanic or Latino | 21 | 20 | 37 | 78
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 5 | 8
  Black or African American | 3 | 3 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 2 | 8
  White | 18 | 19 | 35 | 72
  Other | 2 | 2 | 8 | 12
  Multiple | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  New Zealand | 8 | 5 | 10 | 23
  Canada | 0 | 1 | 3 | 4
  Puerto Rico | 3 | 1 | 5 | 9
  United States | 14 | 18 | 32 | 64
  Israel | 1 | 0 | 0 | 1
  Australia | 3 | 4 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Urinary Albumin-to-creatinine Ratio (ACR)
Description: Data are presented as the geometric mean (GM) of percent change, which is calculated as the geometric mean of the Week 16 ACR to baseline, expressed as percent change from baseline.
Time Frame: Baseline up to Week 16
Population: Intent to Treat Analysis Set
Measure: Geometric Mean (80% Confidence Interval); unit: Geometric Mean of Percent Change
Groups:
- CSL346 (High Dose): Administered as a single intravenous (IV) loading dose followed by subcutaneous (SC) infusions CSL346: VEGF-B antagonist monoclonal antibody
- Placebo: Administered as a single IV loading dose followed by SC infusions Placebo: Normal saline
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose) | Placebo
Number analyzed (Participants) | 28 | 27 | 48
Geometric Mean of Percent Change | 3.2 [-9.79 to 18.05] | 17.7 [2.54 to 35.18] | 5.4 [-3.24 to 14.91]
Statistical Analysis 1: Comparison: CSL346 (Low Dose) vs Placebo; Test type: Superiority; p = 0.485, Mixed Models Repeated Measures Analysis — One-sided p-value; GM % treatment difference (80% CI) = -0.5, 80% CI 2-sided [-14.8 to 16.3] — Data analyzed are log-transformed values of ACR, using MMRM. Comparisons vs. placebo are back-transformed by exponentiation to obtain geometric mean (GM), then expressed as percent treatment difference
Statistical Analysis 2: Comparison: CSL346 (High Dose) vs Placebo; Test type: Superiority; p = 0.750, Mixed Models Repeated Measures Analysis — One-sided p-value; GM % treatment difference (80% CI) = 8.6, 80% CI 2-sided [-7.2 to 27.2] — Data analyzed are log-transformed values of ACR, using MMRM. Comparisons vs. placebo are back-transformed by exponentiation to obtain geometric mean, then expressed as percent treatment difference

2. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Time Frame: Up to 24 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose) | Placebo
Number analyzed (Participants) | 29 | 29 | 54
Participants | 22 | 23 | 32

3. Secondary Outcome: Percentage of Subjects With TEAEs
Time Frame: Up to 24 weeks
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose) | Placebo
Number analyzed (Participants) | 29 | 29 | 54
Percentage of participants | 75.9 | 79.3 | 59.3

4. Secondary Outcome: Number of Subjects With Adverse Events of Special Interest (AESIs)
Description: Data are presented for treatment-emergent AESIs.
Time Frame: Up to 24 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose) | Placebo
Number analyzed (Participants) | 29 | 29 | 54
Participants | 10 | 6 | 13

5. Secondary Outcome: Percentage of Subjects With AESIs
Description: Data are presented for treatment-emergent AESIs.
Time Frame: Up to 24 weeks
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose) | Placebo
Number analyzed (Participants) | 29 | 29 | 54
Percentage of participants | 34.5 | 20.7 | 24.1

6. Secondary Outcome: Observed Value and Mean Change From Baseline in Serum Creatinine
Time Frame: Baseline up to 24 weeks
Population: Intent-to-Treat Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- CSL346 (Low Dose) - Observed; CSL346 (High Dose) - Observed: Administered as a single intravenous (IV) loading dose followed by subcutaneous (SC) infusions.
  CSL346: VEGF-B antagonist monoclonal antibody. Observed value.
- CSL346 (Low Dose) - Change; CSL346 (High Dose) - Change: Administered as a single intravenous (IV) loading dose followed by subcutaneous (SC) infusions.
  CSL346: VEGF-B antagonist monoclonal antibody. Change from Baseline.
- Placebo - Observed: Administered as a single IV loading dose followed by SC infusions. Placebo: Normal saline. Observed value.
- Placebo - Change: Administered as a single IV loading dose followed by SC infusions. Placebo: Normal saline. Change from Baseline.
Arm/Group | CSL346 (Low Dose) - Observed | CSL346 (Low Dose) - Change | CSL346 (High Dose) - Observed | CSL346 (High Dose) - Change | Placebo - Observed | Placebo - Change
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 56 | 56
mg/dL
  Baseline: number analyzed (Participants) | 29 | 0 | 29 | 0 | 54 | 0
  Baseline | 1.273 (0.5502) |  | 1.321 (0.5592) |  | 1.207 (0.5184) |
  Day 8: number analyzed (Participants) | 29 | 29 | 29 | 29 | 53 | 53
  Day 8 | 1.306 (0.5374) | 0.032 (0.1900) | 1.269 (0.5049) | -0.052 (0.1687) | 1.203 (0.5163) | -0.012 (0.1057)
  Day 15: number analyzed (Participants) | 29 | 29 | 28 | 28 | 51 | 51
  Day 15 | 1.306 (0.5229) | 0.032 (0.1634) | 1.218 (0.4838) | -0.079 (0.1838) | 1.234 (0.5318) | 0.013 (0.1080)
  Day 29: number analyzed (Participants) | 29 | 29 | 29 | 29 | 53 | 53
  Day 29 | 1.316 (0.6564) | 0.043 (0.3106) | 1.290 (0.5247) | -0.030 (0.1956) | 1.229 (0.5427) | 0.014 (0.1060)
  Day 57: number analyzed (Participants) | 27 | 27 | 29 | 29 | 48 | 48
  Day 57 | 1.292 (0.6252) | 0.034 (0.1377) | 1.265 (0.5514) | -0.056 (0.1096) | 1.200 (0.4977) | 0.017 (0.1516)
  Day 85: number analyzed (Participants) | 28 | 28 | 27 | 27 | 47 | 47
  Day 85 | 1.285 (0.5621) | 0.025 (0.1725) | 1.226 (0.4711) | -0.050 (0.2002) | 1.251 (0.5409) | 0.030 (0.1371)
  Day 113: number analyzed (Participants) | 28 | 28 | 27 | 27 | 46 | 46
  Day 113 | 1.243 (0.5404) | -0.017 (0.1859) | 1.226 (0.5367) | -0.051 (0.0985) | 1.243 (0.5169) | 0.019 (0.1361)
  Day 169, End of Study: number analyzed (Participants) | 27 | 27 | 27 | 27 | 47 | 47
  Day 169, End of Study | 1.295 (0.6468) | 0.043 (0.2242) | 1.284 (0.5878) | -0.032 (0.1839) | 1.280 (0.5169) | 0.026 (0.1370)

7. Secondary Outcome: Observed Value and Mean Change From Baseline in Estimated Glomerular Filtration Rate (eGFR)
Time Frame: Baseline up to 24 weeks
Population: Intent-to-Treat Analysis Set
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | CSL346 (Low Dose) - Observed | CSL346 (Low Dose) - Change | CSL346 (High Dose) - Observed | CSL346 (High Dose) - Change | Placebo - Observed | Placebo - Change
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 56 | 56
mL/min/1.73 m^2
  Baseline: number analyzed (Participants) | 29 | 0 | 29 | 0 | 54 | 0
  Baseline | 65.38 (25.691) |  | 64.94 (27.960) |  | 71.95 (28.186) |
  Day 8: number analyzed (Participants) | 29 | 29 | 29 | 29 | 53 | 53
  Day 8 | 63.62 (26.433) | -1.77 (9.218) | 66.31 (27.442) | 1.37 (7.400) | 72.57 (28.443) | 1.13 (5.947)
  Day 15: number analyzed (Participants) | 29 | 29 | 28 | 28 | 51 | 51
  Day 15 | 63.02 (25.313) | -2.36 (8.119) | 69.15 (28.175) | 3.09 (9.005) | 70.47 (28.419) | -0.68 (7.230)
  Day 29: number analyzed (Participants) | 29 | 29 | 29 | 29 | 53 | 53
  Day 29 | 65.74 (27.747) | 0.35 (10.433) | 66.12 (28.001) | 1.18 (7.296) | 71.19 (28.935) | -0.26 (5.992)
  Day 57: number analyzed (Participants) | 27 | 27 | 29 | 29 | 48 | 48
  Day 57 | 66.57 (27.555) | -0.26 (7.962) | 67.55 (28.026) | 2.61 (5.496) | 71.98 (28.075) | -0.56 (7.175)
  Day 85: number analyzed (Participants) | 28 | 28 | 27 | 27 | 47 | 47
  Day 85 | 64.33 (24.940) | -1.75 (9.425) | 68.44 (25.535) | 1.00 (7.818) | 69.87 (29.764) | -0.87 (6.522)
  Day 113: number analyzed (Participants) | 28 | 28 | 27 | 27 | 46 | 46
  Day 113 | 66.80 (26.168) | 0.72 (10.277) | 69.77 (27.114) | 2.34 (6.130) | 69.91 (28.493) | -0.32 (6.673)
  Day 169, End of Study: number analyzed (Participants) | 27 | 27 | 27 | 27 | 47 | 47
  Day 169, End of Study | 66.05 (28.012) | -0.56 (11.079) | 67.89 (28.783) | 2.19 (6.456) | 67.70 (28.158) | -1.67 (6.474)

8. Secondary Outcome: Observed Value and Mean Change From Baseline in Systolic Blood Pressure
Time Frame: Baseline up to 24 weeks
Population: Intent-to-Treat Analysis Set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CSL346 (Low Dose) - Observed | CSL346 (Low Dose) - Change | CSL346 (High Dose) - Observed | CSL346 (High Dose) - Change | Placebo - Observed | Placebo - Change
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 56 | 56
mmHg
  Baseline: number analyzed (Participants) | 29 | 0 | 29 | 0 | 54 | 0
  Baseline | 133.4 (10.61) |  | 131.4 (8.63) |  | 133.9 (11.32) |
  Day 8: number analyzed (Participants) | 29 | 29 | 29 | 29 | 53 | 53
  Day 8 | 135.1 (14.21) | 1.7 (12.58) | 133.9 (9.17) | 2.6 (7.37) | 135.7 (11.31) | 1.6 (12.03)
  Day 15: number analyzed (Participants) | 29 | 29 | 28 | 28 | 51 | 51
  Day 15 | 134.4 (16.25) | 1.0 (11.53) | 136.5 (9.10) | 4.4 (8.41) | 135.3 (12.60) | 1.0 (12.82)
  Day 29: number analyzed (Participants) | 29 | 29 | 29 | 29 | 53 | 53
  Day 29 | 135.7 (11.16) | 2.2 (9.02) | 137.7 (10.99) | 6.3 (11.55) | 133.8 (12.04) | -0.2 (12.58)
  Day 57: number analyzed (Participants) | 28 | 28 | 29 | 29 | 49 | 49
  Day 57 | 135.1 (12.75) | 1.0 (12.00) | 134.7 (13.93) | 3.3 (12.44) | 133.1 (13.98) | -0.8 (12.60)
  Day 85: number analyzed (Participants) | 28 | 28 | 27 | 27 | 47 | 47
  Day 85 | 131.5 (13.88) | -2.6 (12.93) | 134.9 (10.69) | 2.3 (10.93) | 135.7 (14.99) | 1.9 (13.15)
  Day 113: number analyzed (Participants) | 27 | 27 | 27 | 27 | 47 | 47
  Day 113 | 136.2 (15.13) | 2.3 (12.23) | 136.9 (8.45) | 4.3 (10.17) | 133.5 (12.93) | 0.4 (12.09)
  Day 169, End of Study: number analyzed (Participants) | 27 | 27 | 27 | 27 | 47 | 47
  Day 169, End of Study | 141.0 (12.00) | 6.4 (10.55) | 132.7 (13.24) | 1.0 (12.20) | 134.6 (15.17) | 1.1 (16.51)

9. Secondary Outcome: Observed Value and Mean Change From Baseline in Diastolic Blood Pressure
Time Frame: Baseline up to 24 weeks
Population: Intent-to-Treat Analysis Set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CSL346 (Low Dose) - Observed | CSL346 (Low Dose) - Change | CSL346 (High Dose) - Observed | CSL346 (High Dose) - Change | Placebo - Observed | Placebo - Change
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 56 | 56
mmHg
  Baseline: number analyzed (Participants) | 29 | 0 | 29 | 0 | 54 | 0
  Baseline | 75.5 (8.55) |  | 73.4 (11.22) |  | 75.5 (8.88) |
  Day 8: number analyzed (Participants) | 29 | 29 | 29 | 29 | 53 | 53
  Day 8 | 76.1 (8.22) | 0.6 (8.95) | 75.4 (11.00) | 2.0 (5.75) | 75.3 (9.73) | -0.3 (7.94)
  Day 15: number analyzed (Participants) | 29 | 29 | 28 | 28 | 51 | 51
  Day 15 | 74.7 (7.34) | -0.9 (7.36) | 77.2 (10.75) | 3.5 (6.52) | 74.4 (8.99) | -1.0 (6.84)
  Day 29: number analyzed (Participants) | 29 | 29 | 29 | 29 | 53 | 53
  Day 29 | 77.2 (6.49) | 1.7 (5.84) | 78.0 (8.58) | 4.5 (8.36) | 75.0 (9.01) | -0.6 (8.17)
  Day 57: number analyzed (Participants) | 28 | 28 | 29 | 29 | 49 | 49
  Day 57 | 76.1 (7.07) | 0.2 (6.90) | 76.8 (9.74) | 3.3 (9.36) | 72.6 (9.96) | -2.5 (7.58)
  Day 85: number analyzed (Participants) | 28 | 28 | 27 | 27 | 47 | 47
  Day 85 | 74.2 (6.57) | -1.7 (7.56) | 77.3 (11.00) | 3.1 (7.67) | 73.3 (10.19) | -1.5 (7.88)
  Day 113: number analyzed (Participants) | 27 | 27 | 27 | 27 | 47 | 47
  Day 113 | 75.7 (7.20) | -0.2 (6.40) | 77.8 (9.94) | 3.6 (7.01) | 73.3 (9.75) | -1.4 (7.33)
  Day 169, End of Study: number analyzed (Participants) | 27 | 27 | 27 | 27 | 47 | 47
  Day 169, End of Study | 77.0 (8.06) | 0.8 (7.83) | 76.0 (11.00) | 2.1 (8.78) | 73.7 (10.88) | -1.0 (8.19)

10. Secondary Outcome: Maximum Concentration (Cmax) After Intravenous (IV) Loading Dose of CSL346 in Serum Samples
Time Frame: Up to 120 minutes after the IV loading dose for CSL346
Population: Pharmacokinetic (PK) Analysis Set
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose)
Number analyzed (Participants) | 29 | 29
ug/mL | 234.26 (671.392) | 182.32 (140.886)

11. Secondary Outcome: Time to Reach Cmax in Serum (Tmax) After IV Loading Dose of CSL346 in Serum Samples
Time Frame: Up to 120 minutes after the IV loading dose for CSL346
Population: PK Analysis Set
Measure: Median (Full Range); unit: Hours
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose)
Number analyzed (Participants) | 29 | 29
Hours | 0.52 [0.0 to 2.0] | 0.55 [0.0 to 2.0]

12. Secondary Outcome: Cmax After First Subcutaneous (SC) Dose of CSL346 in Serum Samples
Time Frame: From Day 1 to Day 29
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose)
Number analyzed (Participants) | 29 | 29
ug/mL | 34.70 (11.405) | 67.88 (29.565)

13. Secondary Outcome: Tmax After First SC Dose of CSL346 in Serum Samples
Time Frame: From Day 1 to Day 29
Population: PK Analysis Set
Measure: Median (Full Range); unit: Hours
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose)
Number analyzed (Participants) | 29 | 29
Hours | 168.05 [119.1 to 671.0] | 167.58 [118.1 to 336.2]

14. Secondary Outcome: Area Under the Concentration-time Curve in First Dosing Interval
Time Frame: From Day 1 to Day 29
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: Hours*ug/mL
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose)
Number analyzed (Participants) | 29 | 29
Hours*ug/mL | 19374.474 (5560.5651) | 37225.571 (13026.7980)

15. Secondary Outcome: Trough Concentration After Each Dose
Time Frame: 29 days after each dose
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose)
Number analyzed (Participants) | 29 | 29
ug/mL
  After first SC dose: number analyzed (Participants) | 29 | 28
  After first SC dose | 15.306 (5.9479) | 28.215 (9.6135)
  After second SC dose: number analyzed (Participants) | 28 | 29
  After second SC dose | 16.686 (7.0049) | 31.541 (9.3408)
  After third SC dose: number analyzed (Participants) | 28 | 27
  After third SC dose | 15.959 (8.1791) | 31.522 (10.1988)
  After fourth SC dose: number analyzed (Participants) | 28 | 27
  After fourth SC dose | 16.225 (6.2157) | 30.544 (10.6822)

16. Secondary Outcome: Number of Subjects Positive for Anti-drug Antibodies
Description: Data are presented for participants who received treatment with CSL346. Any anti-drug antibodies detected in participants who received treatment with Placebo were considered not specific to CSL346 and of no clinical relevance.
Time Frame: Weeks 4, 8, and 16
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose)
Number analyzed (Participants) | 29 | 29
Participants
  Week 4 | 4 | 0
  Week 8: number analyzed (Participants) | 28 | 29
  Week 8 | 4 | 0
  Week 16: number analyzed (Participants) | 28 | 27
  Week 16 | 5 | 0

17. Secondary Outcome: Percentage of Subjects Positive for Anti-drug Antibodies
Description: as for outcome 16
Time Frame: Weeks 4, 8, and 16
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose)
Number analyzed (Participants) | 29 | 29
Percentage of participants
  Week 4 | 13.8 | 0
  Week 8: number analyzed (Participants) | 28 | 29
  Week 8 | 14.3 | 0
  Week 16: number analyzed (Participants) | 28 | 27
  Week 16 | 17.9 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data are presented for the Treatment Period (12 weeks) and the Follow-up Period (up to 12 weeks after the participant's last dose of Investigational Product in the Treatment Period).
Description: Adverse Event data are presented for the Safety Analysis Set.
Arm/Group | CSL346 (Low Dose) | CSL346 (High Dose) | Placebo
All-Cause Mortality (participants affected / at risk) | 1/29 | 1/29 | 0/54
Serious Adverse Events (participants affected / at risk) | 3/29 | 6/29 | 5/54
Other Adverse Events (participants affected / at risk) | 17/29 | 11/29 | 18/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL346 (Low Dose) (N=29) | CSL346 (High Dose) (N=29) | Placebo (N=54)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subdural abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Paroxysmal atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Albuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL346 (Low Dose) (N=29) | CSL346 (High Dose) (N=29) | Placebo (N=54)
COVID-19 (Infections and infestations) | 5 (5) | 3 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (2)
Tooth infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 3 (4) | 1 (1) | 3 (4)
C-reactive protein increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 4 (4)
Albuminuria (Renal and urinary disorders) | 3 (5) | 2 (3) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT04419467/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT04419467/SAP_001.pdf